CLINICAL TRIAL: NCT00950794
Title: Study of Salmeterol (SN408D) for Adult Asthma - Clinical Study of Salmeterol Compared With Hokunalin (Tulobuterol) Tape -
Brief Title: Study of Salmeterol (SN408D) for Adult Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 112376
Record Dates: First submitted 2009-07-30; First posted 2009-08-03 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Asthma; Bronchial Asthma
Keywords: Long acting beta2-agonist
MeSH Terms: conditions — Asthma | interventions — tulobuterol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Hokunalin(tulobuterol) tape (Active Comparator): Hokunalin(tulobuterol) tape: long-acting Beta2-agonist
  Interventions: Drug: Hokunalin (tulobuterol) tape
- Salmeterol(408DP-02) (Experimental): Salmeterol(408DP-02)：long-acting Beta2-agonist
  Interventions: Drug: Salmeterol(SN408D)

INTERVENTIONS:
Drug: Salmeterol(SN408D) — Salmeterol(SN408D)：long-acting Beta2-agonist
  Arms: Salmeterol(408DP-02)
Drug: Hokunalin (tulobuterol) tape — Hokunalin (tulobuterol) tape:long-acting Beta2-agonist
  Arms: Hokunalin(tulobuterol) tape

SUMMARY:
To demonstrate the efficacy (non-inferiority) of Salmeterol 50mcg bid (100mcg/day), compared with Hokunalin (tulobuterol) tape 2mg once a day, in terms of improvement in pulmonary function (peak expiratory flow: PEF) in a randomized, double-blind, parallel-group comparative study in adult patients with bronchial asthma on ICS 400mcg/day of FP equivalent.

DETAILED DESCRIPTION:
Primary To demonstrate the efficacy (non-inferiority) of Salmeterol 50mcg bid (100mcg/day), compared with Hokunalin (tulobuterol) tape 2mg once a day, in terms of improvement in pulmonary function (peak expiratory flow: PEF) in a randomized, double-blind, parallel-group comparative study in adult patients with bronchial asthma on ICS 400mcg/day of FP equivalent.

Secondary

* To evaluate the efficacy of Salmeterol , compared with Hokunalin (tulobuterol) tape in terms of asthma symptoms recorded in the asthma diary.
* To evaluate the safety of Serevent compared with Hokunalin (tulobuterol) tape.

ELIGIBILITY:
Inclusion Criteria:

* For entry into run-in period (Visit 1)

A subject will be considered eligible for inclusion in this study only if all of the following criteria apply:

1. Males or females aged >= 15 years at the time of giving informed consent.
2. Subjects who are able to give a written informed consent to participation in the study.

   However, if a subject is aged < 20 years at the time of giving informed consent, a written informed consent should be obtained from the subject and his/her legally acceptable representative.
3. Outpatients.
4. Subjects who had been diagnosed as asthma at least 6 months prior to Visit 1.
5. Subjects who have been receiving ICS 400mcg/day of FP equivalent for at least 8 weeks prior to Visit 1.

   * For entry into the treatment period (Visit 2)

A subject will be considered eligible for entering the treatment period only if he/she completes the run-in period and meets all of the following criteria:

1. Subjects who meet both of the following criteria in terms of pulmonary function.

   * Has a mean morning PEF during the last 7 days (at least 4 days) prior to Visit 2 is >= 40% of the predicted value.
   * Has at least 2 days with a diurnal variation in PEF of >= 15% during the run-in period, or had been confirmed and recorded reversibility of >= 15% using rapid-acting inhaled beta2 agonists within 3 months prior to Visit 1 (including Visit 1).
2. Subjects who have >= 70 % compliance with asthma medication during the run-in period.
3. Subjects who were able to measure peak flows correctly during the run-in period, in the investigator's/subinvestigator's judgment.
4. Subjects who were able to keep the asthma diary correctly during the run-in period, in the investigator's/subinvestigator's judgment.

Exclusion Criteria:

* A subject will not be eligible for inclusion in this study if any of the following criteria apply at Visit 1 or Visit 2:

  1. Subjects who have received injected steroids, injected ACTH, or oral steroids within four weeks of Visit1 or during run-in period.
  2. Subjects who have received xanthines (oral, injected, suppository), beta2 agonists other than rescue medication (rapid-acting inhaled beta2 agonists), or inhaled anti-cholinergics during the run-in period.
  3. Subjects with respiratory disease other than asthma (e.g., chronic bronchitis, emphysema, bronchiectasis, pulmonary fibrosis, lung cancer, sarcoidosis, and old tuberculosis) which, in the judgment of the investigator/subinvestigator, are likely to affect efficacy evaluation.
  4. Subjects with uncontrollable diabetes mellitus, hypertension, heart disease, or hyperthyroidism, who are inappropriate for this study in the judgement of the investigator/sub investigator.
  5. Subjects who are unsuitable for this study in the judgment of the investigator/subinvestigator based on 12-lead ECG findings at Visit 1.
  6. Subjects who are regularly using medications containing the following ingredients:

     beta-blockers, alpha/beta-blockers
  7. Subjects who have received immunosuppressive medications excluding Tacrolimus ointment.
  8. Subjects who are receiving catecholamines.
  9. Subjects with atopic dermatitis who are inappropriate for this study in the judgment of the investigator/subinvestigator.
  10. Subjects who had or are suspected to have had hypersensitivity to any of the investigational products.
  11. Subjects who received the last dose of other investigational drugs in the past 30 days.
  12. Subject who are currently pregnant, possibly pregnant, lactating or willing to become pregnant during the study period.
  13. Subjects who consume alcohol or drugs excessively the opinion of the investigator/subinvestigator.
  14. Subjects who are judged by the investigator/subinvestigator to have Step 4 asthma (severe persistent), referring to "GINA2002" and "J-GL2003"．
  15. Subjects who are judged by the investigator/subinvestigator to be inappropriate for this study for any other reasons.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2003-09; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Change in morning PEF | 8 week

SECONDARY OUTCOMES:
Use of short acting beta agonist | 8 week
Adverse event | 8 week
Evening PEF | 8 week
Symptom score | 8 week

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline